CLINICAL TRIAL: NCT01265758
Title: OPTIMIZING DIAGNOSTICS AND THERAPY OF ARRHYTHMIA AND SYNCOPE EVENTS USING INTELLIGENT TELEMETRIC SOLUTIONS - Evaluation of Arrhythmia Diagnostics in Adults
Brief Title: Telemetric Arrhythmia Diagnosis in Adults
Acronym: TELEMARC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Prof Lukasz Szumowski, Institute of Cardiology, Warsaw Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UDAPOIG.01.03.01-00-068/09-00A
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Atrial fibrillation; Cardiac arrhythmia; ECG; Telemonitoring; Telemetry; Holter
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemetric ECG monitoring (Experimental): Telemetric 14-days Full Disclosure ECG recording.
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.
- Standard 24-hours Holter ECG recording (Active Comparator): Standard 24-hours Holter ECG recording repeated 3 times unless arrhythmia is diagnosed earlier.
  Interventions: Device: Prolonged telemetric Full Disclosure ECG recording.

INTERVENTIONS:
Device: Prolonged telemetric Full Disclosure ECG recording. — Continuous Full Disclosure Telemetric ECG monitoring lasting 14 days
  Other Names: Medicalgorithmics, PocketECG

SUMMARY:
The purpose of this study is to assess efficacy of prolonged Full Disclosure electrocardiogram (ECG) monitoring and signal analysis using advanced telemetric technology in comparison with a standard Holter ECG recording and an Event Holter recording to diagnose cardiac arrhythmia.

DETAILED DESCRIPTION:
Irregular and/or rapid beating of the heart called heart palpitations can occur in individuals without heart disease and the reasons for their palpitations are unknown. Together with heart palpitations silent arrhythmia may be present that could lead to serious complications (eg. stroke). In others, palpitations result from heart rhythm disturbances, sometimes life threatening. Standard diagnostic methods such as 24 hours Holter ECG monitoring or Event Holter do not guarantee early diagnosis of the arrhythmia. Prolonged heart rhythm recording and analysis using an automatic full disclosure telemetric device increase probability of arrhythmia diagnosis and early administration of applicable treatment. Study patients will be diagnosed using standard Holter ECG monitoring and 14 days telemetric full disclosure ECG monitoring. The full disclosure signal will be subsequently analyzed in the Event Monitoring mode by an independent consultant. Efficacy of Telemetric Monitoring in diagnosis of cardiac arrhythmia will be assessed in comparison with the standard Holter monitoring and Event Monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age - between 18 and 80 years old
* History of symptoms potentially caused by arrhythmia
* Symptoms occuring at least monthly
* Patient informed consent
* Declarative and feasible compliance (patient understands basic instructions regarding device use)

Exclusion Criteria:

* Evidence of previously recorded arrhythmia
* Inability to comply with the study protocol
* Lack of patient cooperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Recording of symptomatic or life threatening arrhythmia event | 14 days
  ECG monitoring is conducted until occurrence of symptomatic arrhythmia or life threatening arrhythmia but not longer than 14 days. Patients in the control group will have standard ECG Holter monitoring repeated 3 times unless arrhythmia is diagnosed earlier.

SECONDARY OUTCOMES:
Quality of Life questionnaire and European Heart Rhythm Association (EHRA) scale assessment against evidence of cardiac arrhythmia occurrence. | 14 days
  Verification of patient self assessment based on the Quality of Life questionnaire and European Heart Rhythm Association (EHRA) scale against evidence of cardiac arrhythmia occurrence.
Silent (asymptomatic) arrhythmia events incidence detection assessment | 14 days
  Evaluation of silent (asymptomatic) arrhythmia events incidence which potentially could cause serious complications
  1. Atrial fibrillation
  2. Atrial flutter
  3. Atrial Tachycardia
  4. Ventricular tachycardia
Evaluation of stroke and bleeding risk factors incidence | 14 days
  Evaluation of stroke and bleeding risk factors incidence based on scores proposed in the European Society of Cardiology (ESC) guidelines: CHADS2VASC2 and HAS-BLED.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz J Szumowski, MD, PhD, Study Chair — National Institute of Cardiology, Warsaw, Poland
Locations (2):
- Poland (2):
  - The Medical University of Gdańsk, Gdansk
  - Institute of Cardiology, Warsaw